CLINICAL TRIAL: NCT04923672
Title: Evaluation of the Feasibility of Wearable Technology-Guided Exercise Preconditioning to Accelerate Return to Function After Cancer Surgery
Brief Title: Exercise Preconditioning with Cancer Surgeries
Acronym: ExPre 01
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Company providing the computer application for exercise intervention suddenly closed for business
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Traci Hedrick, MD, Associate Professor, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 210103
Record Dates: First submitted 2021-06-07; First posted 2021-06-11 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Colorectal Cancer; Hepatobiliary Cancer; Gynecologic Cancer
Keywords: Prehabilitation; Exercise; Physical activity
MeSH Terms: conditions — Colorectal Neoplasms; Motor Activity | interventions — High-Intensity Interval Training

STUDY DESIGN:
Intervention Model Description: Randomization to either control group or one of two exercise groups: moderate continuous or high intensity interval training
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control group (No Intervention): Participants will be asked to wear an Apple watch through about 30 days after surgery and will be asked to maintain their current activity level.
- Moderate continuous training group (Active Comparator): Apple watch and a smartphone application
  Increase activity to 5 days a week, 40 minutes a day of continuous moderate intensity exercise prior to surgery.
  Interventions: Behavioral: Moderate continuous exercise
- High intensity interval training group (Active Comparator): Apple watch and a smartphone application
  Increase activity to 5 days a week, 40 minutes a day of intervals of high and moderate intensity exercise prior to surgery.
  Interventions: Behavioral: High intensity interval exercise

INTERVENTIONS:
Behavioral: Moderate continuous exercise — Participants will be asked to wear an Apple watch and use a smartphone application to help increase their activity to 5 days a week, about 40 minutes a day of continuous moderate intensity exercise prior to surgery. They will be asked to continue wearing the watch through about 30 days after surgery.
  Arms: Moderate continuous training group
Behavioral: High intensity interval exercise — Participants will be asked to wear an Apple watch and use a smartphone application to help increase their activity to 5 days a week, about 40 minutes a day of intervals of high and moderate intensity exercise prior to surgery. They will be asked to continue wearing the watch through about 30 days after surgery.
  Arms: High intensity interval training group

SUMMARY:
Studies have shown that people who are more physically fit prior to surgery do better after surgery. For this reason, it may be helpful for people who are going to have abdominal surgery for cancer to exercise before surgery to increase fitness. In this study, patients will be assigned to either maintain their current activity, or increase activity to 5 days a week, 40 minutes per day, of either continuous moderate activity or intervals of moderate and vigorous activity (three groups). All participants will wear an Apple watch, and participants in the exercise groups will use a smartphone application to get feedback on activity and encouragement to reach activity goals.

DETAILED DESCRIPTION:
Research indicates that people who have better physical fitness at the time of surgery have a better chance of surviving the surgery and returning to normal function. An exercise intervention in the 3+ weeks before surgery (after the decision that surgery is necessary) may help people who are going to have abdominal surgery for cancer increase fitness prior to surgery. Devices that track physical activity, like smartwatches or Fitbits, allow the wearer to get feedback on physical activity information like steps taken, distance traveled, time in light, moderate or vigorous activity and on heart rate. Having this information and using a smartphone application designed to increase physical activity may help patients increase physical activity and thereby fitness, prior to abdominal surgery for cancer.

The main goal of this project is to test two physical activity interventions and also a "control group" to make sure that participants can do the interventions and to see whether there are changes in activity and fitness in each group:

1. Control group - maintain current activity
2. Moderate continuous activity group - increase activity to 5 days a week, 40 minutes per day, of continuous moderate activity
3. High Intensity Interval Training group - increase activity to 5 days a week, 40 minutes per day, of intervals of moderate and vigorous activity

All participants will wear an Apple watch, and participants in the exercise groups will use a smartphone application to get feedback on activity and encouragement to reach activity goals.

Optional: Participants will also be asked to provide a small amount of blood for research purposes.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥ 18 years of age) patients undergoing elective abdominal oncologic resection of a confirmed or potential colorectal, hepatobiliary, or gynecologic neoplasm.
* Study participants must be able to provide written informed consent and authorization.
* Study participants must be able to understand written and verbal English, as well as to be able to communicate in English.
* Study participants must have an Apple iphone to use during the study period

Exclusion Criteria:

* Any patient unable and/or unwilling to cooperate with all study protocols.
* Patients who require an assist device (walker) for ambulation.
* Patients that indicate they did at least 3 days of vigorous intensity activity in the previous 7 days OR any combination of walking, moderate-intensity or vigorous-intensity in all of the last 7 days totaling at least 18 and a half hours
* Recent history of cardiac disease (within 3 months of registration) that would preclude vigorous exercise
* Individuals with end stage renal disease currently on dialysis
* Individuals with a history of liver failure as evidenced by AST, ALT or Alkaline Phosphatase ≥ 3x upper limit of normal
* Individuals with uncontrolled hypertension
* Women who are breastfeeding or pregnant
* American Society of Anesthesiologists Physical Status score ≥ 4
* Any patient that needs further cardiac evaluation per ACC/AHA perioperative criteria
* Surgery scheduled < 3 weeks of study registration (precluding time to participate in exercise regimen)
* Any patient who currently uses a fitness tracker or heart rate monitoring-capable device to guide exercise
* Patient indicates a lack of familiarity or discomfort with using a smartphone
* If participation is not in the best interest of the patient, in the opinion of the treating investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-02-20 (Actual); Primary Completion 2024-09-12 (Actual); Study Completion 2024-09-12 (Actual)

PRIMARY OUTCOMES:
Steps per day | Baseline through the 1 day visit prior to surgery
  Change in average steps per day measured at baseline and at the time of surgery

SECONDARY OUTCOMES:
Enrollment rate | During participant accrual, estimated to take about 12 months
  Number of participants enrolled per month
Compliance with EXi smartphone application | From baseline through 1 day visit just prior to surgery
  To assess feasibility of the intervention
Compliance with exercise intervention, including percentage of exercise goals reached | From baseline through 1 day visit just prior to surgery
  To assess feasibility of the intervention
Completion/Dropout rate | From baseline through about 30 days after surgery
  To assess feasibility of the intervention
Percentage of time wearing Apple Watch | From baseline through about 30 days after surgery
  To assess feasibility of the intervention
Health-related quality of life | Baseline and 1 day of surgery
  As measured by PROMIS Global Health Scale
Pain intensity | Baseline and 1 day of surgery
  As measured by PROMIS Pain intensity
Pain interference | Baseline and 1 day of surgery
  As measured by PROMIS Pain interference
Physical activity level by self report | Baseline and 1 day of surgery
  As measured by the International Physical Activity Questionnaire
Surgical complications | 30 days after surgery
  Based on review of medical records
Length of hospital stay (in days) following surgery | Up to 30 days following surgery
  Days participant stayed in hospital following surgery date
Steps per day | From baseline through 30 days after surgery
  Measured by Apple Watch
Fitness level | Baseline, 1 day prior to surgery, and 30, 90, and 180 days following surgery
  As measured by 6 minute walk test

CONTACTS AND LOCATIONS:
Overall Officials: Traci Hedrick, MD, Principal Investigator — UVA
Locations (1):
- UVA Health System, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No